CLINICAL TRIAL: NCT01020110
Title: Human Umbilical Vein Endothelial Cells (HUVEC)-Perfusion
Brief Title: Study in an Ex-vivo Thrombosis Model With Human Umbilical Vein Endothelial Cells (HUVEC)-Perfusion
Acronym: HUVEC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ghazaleh Gouya, Dr., Medical University of Vienna
Other Study IDs: HUVEC-Version1
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Thrombosis; Thrombus Formation; Thrombus Stability
Keywords: perfusion chamber; thrombus D-Dimer; HUVEC
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — supernatant of plasmin degraded thrombus including fibrin monomers
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of fibrin and platelet deposition on a human umbilical endothelial cell surface in perfusion chamber experiments using human whole blood.

Open-label, non interventional study Perfusion chamber experiment will be performed in 30 healthy patients. The Impact of different pH-solutions on thrombus lysis will be evaluated in an in-vitro second step

Outcome:

D-Dimer content of the thrombus reflecting the size of the thrombus.

DETAILED DESCRIPTION:
All Subjects will have two perfusion chamber experiment as follow with an estimated maximum of blood loss of 165ml:

Before blood perfusion, perfuse the system including the chambers with human umbilical vein endothelial cell coated glass slides (HUVEC), with sodium chloride (NaCl) (0.9%), to ensure no leaks and to remove all air bubbles.

Blood is drawn from a vein in the arm with a Surflo® Winged Infusion Set, 19G (Terumo Europe, Leuven, Belgium) with a pump (Masterflex® L/S™, Cole-Parmer Instrument Company, Vernon Hills, Illinois, USA). Five mL of blood is discarded before each perfusion.

Three in serial placed flow chambers (with HUVEC) heated to 37°C are used. They are made of a Plexiglas block through which a cylindrical hole of 0.2 cm in diameter is machined. The aorta pieces are perfused at 10 mL/min for 5 minutes, followed by a 30 seconds perfusion with NaCl (0.9%).

The plasmin degraded thrombus D-Dimer content will be further evaluated under different conditions (different pH solutions).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Use of any medication
* Current diseases
* Anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
D-Dimer content of the plasmin degraded thrombus | Assessment will follow after all perfusion chamber experiments (1 week)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna- Dept. of Clinical Pharmacology, Vienna, Austria